CLINICAL TRIAL: NCT03921190
Title: Should Maxillary Buccal Infiltration Anesthesia be Given in a Closed Mouth Technique? - a Clinical Study
Brief Title: Should Maxillary Buccal Infiltration Anesthesia be Given in a Closed Mouth Technique?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Ahmad El-Ma'aita, Principal investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1012018/3686
Record Dates: First submitted 2019-03-30; First posted 2019-04-19 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia, Local; Pain Control
Keywords: Buccal infiltration anesthesia; Discomfort
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Providing dental local anesthesia (maxillary buccal infiltration) using two techniques; open-mouth and closed-mouth
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-mouth (Active Comparator): Patients receiving maxillary buccal infiltration anesthesia (MBIA) with their mouth wide open
  Interventions: Procedure: Local anesthesia
- Closed-mouth (Experimental): Patients receiving MBIA using a closed-mouth technique
  Interventions: Procedure: Local anesthesia

INTERVENTIONS:
Procedure: Local anesthesia — Patients scheduled for a dental procedure that requires local anesthesia will be given the injection using two 2 techniques; an open-mouth and closed-mouth techniques

SUMMARY:
To study the patients' and dentists' perception of receiving/ administering maxillary buccal infiltration anesthesia using an open or closed mouth techniques

DETAILED DESCRIPTION:
Background: Local anesthesia is an essential part of dentistry. The most commonly used technique to anesthetise maxillary posterior teeth is buccal infiltration with a local anesthetic agent. The technique described in the literature focuses on the location of injection, the direction of the needle insertion in relation to the root apex, the direction of needle bevel in relation to the cortical bone plate, the size of needle and the type and amount of the local anesthetic agent used. However, there is no mention to whether the patient should open their mouth or maintain their teeth in intercuspation during the injection procedure.

Aims: This research aims to a) compare two techniques of injection (open and closed-mouth techniques) in terms of the discomfort experienced by patients during the injection procedure and b) evaluate the dentists' preference in performing either of the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (16 years old and older)
* Healthy (American Society of Anaesthesiologists (ASA) category I or II)
* A maxillary posterior tooth (excluding third molars) referred for root canal treatment and diagnosed with irreversible pulpitis and normal apical tissues

Exclusion Criteria:

* Psychological disorders
* Intraoral soft tissue abnormalities
* necrotic pulp with/ without apical pathology
* tenderness to palpation and/or percussion
* The use of analgesics in the preceding 12 hours before the appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad El-Ma'aita, PhD, Principal Investigator — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Select One, Jordan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-mouth | Closed-mouth
Started | 56 | 64
Completed | 56 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-mouth | Closed-mouth | Total
Number analyzed (Participants) | 56 | 64 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (14.7) | 39.6 (14.9) | 39.3 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 38 | 69
  Male | 25 | 26 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Perception
Description: Pain perception during local anesthesia injection on a standard 100mm visual analogue scale (VAS) where zero indicates no pain at all and 100 indicates intolerable pain/ worst imagined pain (scale attached in the protocol section). The average scores were calculated for each group and compared. Higher values indicated higher pain/ discomfort experienced during the injection procedure.
Time Frame: 5 minutes after receiving the injection
Population: Study participants
Measure: Mean (Standard Deviation); unit: millimeters on a visual analogue scale
Arm/Group | Open-mouth | Closed-mouth
Number analyzed (Participants) | 56 | 64
millimeters on a visual analogue scale | 32.6 (15.8) | 25 (14)

2. Secondary Outcome: Dentist Perception of Visibility During Anesthesia Injection
Description: Participating dentists were asked to rate the visibility of injection site and ease of cheek retraction during injection on a standard 100mm visual analogue scale where 100 indicates the best possible visibility/ easiest cheek retraction and 0 means no visibility at all/ most difficult cheek retraction. The mean scores were compared between the 2 groups using independent t-test.
Time Frame: 30-60 days
Population: Patients receiving maxillary buccal infiltration anesthesia
Measure: Mean (Standard Deviation); unit: millimeters on a visual analogue scale
Arm/Group | Open-mouth | Closed-mouth
Number analyzed (Participants) | 233 | 236
millimeters on a visual analogue scale
  Visibility during injection | 68.1 (17.1) | 82.6 (14.3)
  Ease of cheek retraction | 64.9 (20.1) | 83.2 (12.7)

3. Secondary Outcome: Dentist Preference of Performing One of the Two Techniques of Maxillary Buccal Infiltration; Open-mouth or Closed-mouth
Description: Number of dentists preferring each technique
Time Frame: 3-60 days
Population: Practicing dentists performing local anesthesia
Measure: Count of Participants; unit: Participants
Groups:
- Open-mouth: Number of dentists who preferred the open-mouth technique for maxillary buccal infiltration anesthesia
- Closed-mouth: Number of dentists who preferred the closed-mouth technique for maxillary buccal infiltration anesthesia
Arm/Group | Open-mouth | Closed-mouth
Number analyzed (Participants) | 48 | 48
Participants | 3 | 38

ADVERSE EVENTS:
Time Frame: Up to 1 hour after injection
Arm/Group | Open-mouth | Closed-mouth
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/64
Other Adverse Events (participants affected / at risk) | 0/56 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03921190/Prot_SAP_000.pdf